Microcurrent Dressing to Treat Infections, Before, During and After Surgery

NCT03156543

2018-01-05

# **Evaluation of a Microcurrent Dressing for Prophylaxis Against Perioperative Prosthetic Joint Infection**

PI: Bruce Miller, MD

Co-Is: Asheesh Bedi, Margaret Paulauski, Brian Downie, Tristan Maerz

Study personnel: Elizabeth Sibilsky Enselman, Jaimee Gauthier

## Lay Explanation

The purpose of the study is to evaluate the efficacy of a microcurrent dressing in eliminating certain bacteria that is found on our skin, thus it would reduce the risk of shoulder infections.

Deep periprosthetic infection following total joint arthroplasty is a major complication. Although it only occurs in a small percentage of patients ( $\sim$ 1%), it results in substantial complications and a decline in functional outcome. A two stage revision and exchange is commonly required in order to clear the infection and provide the best opportunity for prosthetic replantation.

Propionibacterium Acnes is bacteria that are found in hair follicles, sebaceous glands, and moist areas of the shoulder and armpit. Because of its low virulence, infections caused by P. acnes typically have a low-grade, slow course, with shoulder pain often the only presenting symptoms after prosthetic replacement. P. acnes is particularly challenging to both diagnose and to eradicate, and is a substantial source of low quality and functional outcomes with shoulder arthroplasty.

JumpStart<sup>TM</sup> is a wireless, advanced microcurrent generating dressing used for the management of surgical incision sites. Microcell batteries made of silver and zinc, generate an electrical current when activated by conductive fluids, such as saline, hydrogel or bodily fluids from a wound. These microcells create low voltage electrical fields to stimulate the surrounding area and to provide antimicrobial protection to assist with wound healing. JumpStart has demonstrated superior broad spectrum bactericidal activity of a wound dressing against antibiotic-resistant strains of wound isolates within 24 hours.



The use of JumpStart as a prophylactic preoperative and post-operative dressing to alter the skin flora and thereby decrease the risk of prosthetic infection has not been investigated to-date. Given the morbidity of a prosthetic infection, this would be a remarkably valuable intervention for any joint replacement procedure.

## **Background**

Deep periprosthetic infection following total joint arthroplasty is a major complication. Although it only occurs in a small percentage of patients (~1%), it results in substantial morbidity and a decline in functional outcome. A two stage revision and exchange is commonly required in order to clear the infection and provide the best opportunity for prosthetic replantation. Following removal of the infected components, a minimum course of six weeks of parenteral antibiotics is given and resolution of the infection confirmed through the ESR, CRP, and repeated aspiration of the joint. In most instances a temporary spacer of antibiotic-loaded cement is inserted at the first stage and removed at the second operation.

Propionibacterium Acnes is a gram-positive, non-spore-forming, anaerobic bacillus found in lipid-rich areas, including hair follicles, sebaceous glands, and moist areas of the shoulder and axilla. Because of its low virulence, infections caused by P. acnes typically have a low-grade, indolent course, with shoulder pain often the only presenting symptoms after prosthetic replacement. P. acnes is particularly challenging to both diagnose and to eradicate, and is a substantial source of morbidity with shoulder arthroplasty.

JumpStart<sup>TM</sup> is a wireless, advanced microcurrent generating, dressing used for the management of surgical incision sites. Microcell batteries made of silver and zinc, generate an electrical current when activated by conductive fluids, such as saline, hydrogel or wound exudate. These microcells create low voltage electrical fields to stimulate the surrounding area and to provide antimicrobial protection to assist with wound healing. JumpStart has

demonstrated superior broad spectrum bactericidal activity of a wound dressing against antibiotic-resistant strains of wound isolates within 24 hours.

The use of JumpStart as a prophylactic preoperative dressing to alter the skin flora and thereby decrease the risk of prosthetic infection has not been investigated to-date. Given the morbidity of a prosthetic infection, this would be a remarkably valuable intervention for any joint replacement procedure.

Due to lower than expected accrual, the addition of arthroscopic shoulder surgery patients will still allow the study of the JumpStart dressing and the efficacy of eliminating P. acnes in a board patient population.

Objective: To evaluate the efficacy of a microcurrent dressing in eliminating P. acnes skin colonization and thereby reduce the risk of perioperative prosthetic shoulder infection.

*Overall Study Design.* This is a prospective cohort study of patients that are scheduled to have a total or reverse shoulder arthroplasty or arthroscopic shoulder surgery. There will be two groups for this study. Both groups will follow the same timeline below.

Group A: With the exception of the preoperative JumpStart dressing and cultures for assessment of P. acnes which will be paid for with department funds the study does not deviate from the standard of care typically provided to patients seeking treatment for a total or reverse shoulder arthroplasty or arthroscopic shoulder surgery within the University of Michigan Health System, and is in line with national and international standards of care.

Group B: With the exception of the preoperative and postoperative JumpStart dressing and cultures for assessment of P. acnes which will be paid for with department funds the study does not deviate from the standard of care typically provided to patients seeking treatment for a total or reverse shoulder or arthroscopic shoulder surgery arthroplasty within the University of Michigan Health System, and is in line with national and international standards of care.

An overview of the timeline of study visits is presented in Table 1.

| Study Visit | Approx. Time<br>from Initial<br>Visit | Measures Performed |
|---|---|---|
| Study Enrollment Visit/ H&P Visit | -4wks to -<br>1wks prior to<br>surgery | Consent |
| Research Visit | -2d | Placement of JumpStart dressing, skin culture |
| Surgery | 0 | Skin culture and biopsy; Group B Postoperative JumpStart dressing applied |
| Post-op Research Visit | 7 days | Removal of dressing for both groups, images of incision and reapplication of |

10-14d

Skin culture, images of incision

**Table 1.** Timeline of study visits and measures performed in study.

Subject Selection and Recruitment. The inclusion criteria will be strictly limited to total or reverse shoulder arthroplasty or arthroscopic shoulder surgery. Exclusion criteria- under the age of 18, revision shoulder arthroplasty patients, sensitivity or allergy to sliver or zinc or latex.

Patients will be recruited from clinic in Orthopaedic Surgery. Patients who seek treatment and who are deemed to be potential candidates for a total or reverse shoulder arthroplasty or arthroscopic shoulder surgery will be approached to participate in the research study.

JunpStart Dressing. Groups A and B will have the dressing applied 2 days prior to surgery by a member of the research team. Sterile saline will be used to moisten the dressing. Group B then will have the dressing again applied at the conclusion of surgery. This will be done using routine UM surgical OR protocols. Both groups will report for a research visit 7 days after surgery for a dressing check. Group B will have another JumpStart dressing reapplied until they report back for their first PO visit 10-14 days after surgery. Group A will have the same type of dressing reapplied that was placed on after surgery.

Measurement of P.Acnes. Twenty patients scheduled for total or reverse shoulder arthroplasty or arthroscopic shoulder surgery will have a topical skin culture in duplicate at the site of the deltopectoral incision 48 hours before the surgical procedure. Then a Jumpstart dressing will be applied to the deltopectoral incision site and left in place until intraoperative preparation and draping for the surgical procedure. Prior to preparation with chlorhexidine, a topical skin culture will be taken in duplicate. The skin will then be prepared for surgery in the standard fashion, and the deltopectoral incision will be made. A small biopsy from the edge will be taken for deep tissue culture and evaluation.

All topical and deep tissue specimens will be cultured for aerobic and anaerobic cultures, including specific culture for Propionibacterium Acnes. The type and number of colony forming units (CFU) will be recorded.

Chart Review. Patients' chart will be monitored for clinical outcomes related to shoulder surgery and any cases of acute, subacute, or chronic prosthetic infection and will be recorded for a minimum of a year postoperatively.

*Images.* At 7 and then again 10-14 day postoperatively, the wound will be inspected and images will be obtained to evaluate cosmesis and apposition. Care will be taken to protect subject's privacy.

**Group Assignment.** Subjects will be randomly assigned to either group A or B. There will be a 50% chance of being assigned to either group.

#### Risks

## The risks associated with the research study include:

<u>Skin Cultures and Biopsy:</u> There are no risks related to the skin cultures. These are taken topically. The skin biopsy will be taken prior to incision closure and should not cause extra scaring as it will be taken form the margin of the incision.

<u>JumpStart Dressing:</u> Should not be use on individuals with sensitivity or allergy to silver, zinc, latex. MRI Non Compatible: Neither MRI Safe nor MRI Compatible and should not be used in conjunction with MRI systems. Frequent or prolonged use of this product may result in permanent discoloration of the skin (i.e. argyria). The use of adhesive dressings on fragile or sensitive skin may pose a risk of skin damage upon removal of the dressing. The patient should stop using the dressing and consult a physician if allergy, irritation, increased pain, maceration or any irregular skin discoloration occurs.

### **Confidentiality:**

There is a small risk of breach of confidentiality. Your research data will not leave the University of Michigan medical campus (Ann Arbor, MI). Data and images will be retained until data related to the research is published at which time all the materials will be destroyed.

As with any research study, there may be additional risks that are unknown or unexpected.

#### **Data Safety Monitoring Plan**

The risk level indicated for this study is no more than minimal risk. All study team members including PI, Co-Is, study coordinators, and research assistants will obtain informed consent, and will provide study information and instructions to the subjects beyond what is included in the informed consent document, and will collect and record study data.

Adverse events will be reported to the IRB using the standard IRBMED AE reporting timetable, utilizing the generalized AE grading scale:

- 0 No adverse event
- 1 Mild AE: No treatment needed
- 2 Moderate AE: Resolved with treatment
- 3 Severe AE: Inability to carry on normal activities, required professional medical attention
- 4 Life-threatening or disabling AE
- 5 Fatal AE

Serious Adverse Events (SAEs) will be categorized according to the following FDA definition:

- Death
- A life-threatening adverse drug experience
- Inpatient hospitalization or prolongation of existing hospitalization
- A persistent or significant disability/incapacity

- A congenital anomaly/birth defect
- Important medical events that may not result in death, be life-threatening, or require hospitalization may be considered a serious adverse drug experience when, based upon appropriate medical judgment, they may jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the outcomes listed in this definition.

The PI and/or Co-I will determine the attribution/relatedness for each AE in the following manner:

- Definitely related
- Probably related
- Possibly related
- Unlikely to be related
- Definitely not related

The expectedness will be assigned for each AE according to the following definitions: <u>Unexpected adverse events</u> (i.e., has NOT been addressed or described in one or more of the following: Informed consent document(s) for this study, IRB application for this study, protocol or procedures for this study, published literature, other documentation)

**Expected adverse events** (i.e., has been addressed or described in one or more of the following: Informed consent document(s) for this study, IRB application for this study, protocol or procedures for this study, published literature, other documentation, or characteristics of the study population)

The frequency with which the study team will conduct scheduled assessments of study recruitment, data integrity and quality, adverse events, withdrawals, and compliance with protocol plan will be on a quarterly basis because this is a minimal risk study. No additional monitoring is required – the nature, size, and complexity of this study does not require additional safety monitoring to that provided by the IRB. Monitoring reports will be provided to the IRB.

#### **Related Literature:**

- 1. Coste JS, Reig S, Trojani C, Berg M, Walch G, Boileau P. The management of infection in arthroplasty of the shoulder. J Bone Joint Surg Br. 2004 Jan;86(1):65-9.
- 2. Sperling JW, Hawkins RJ, Walch G, Mahoney AP, Zuckerman JD. Complications in total shoulder arthroplasty. Instr Course Lect. 2013;62:135-41.
- 3. Sperling JW, Kozak TK, Hanssen AD, Cofield RH. Infection after shoulder arthroplasty. Clin Orthop Relat Res. 2001 Jan;382:206-16.
- 4. Levy PY, Fenollar F, Stein A, Borrione F, Cohen E, Lebail B, Raoult D. Propionibacterium acnes postoperative shoulder arthritis: an emerging clinical entity. Clin Infect Dis. 2008 Jun 15;46(12):1884-6.
- 5. Pottinger P, Butler-Wu S, Neradilek MB, Merritt A, Bertelsen A, Jette JL, Warme WJ, Matsen FA 3rd. Prognostic factors for bacterial cultures positive for Propionibacterium acnes and other organisms in a large series of revision shoulder arthroplasties performed for stiffness, pain, or loosening. J Bone Joint Surg Am. 2012 Nov 21;94(22):2075-83.

- 6. Grosso MJ, Frangiamore SJ, Saleh A, Kovac MF, Hayashi R, Ricchetti ET, Bauer TW, Iannotti JP. Poor utility of serum interleukin-6 levels to predict indolent periprosthetic shoulder infections. J Shoulder Elbow Surg. 2014 Sep;23(9):1277-81. Epub 2014 Apr 13.
- 7. Foruria AM, Fox TJ, Sperling JW, Cofield RH. Clinical meaning of unexpected positive cultures (UPC) in revision shoulder arthroplasty. J Shoulder Elbow Surg. 2013 May;22(5):620-7. Epub 2012 Sep 13.
- 8. Strickland JP, Sperling JW, Cofield RH. The results of two-stage re-implantation for infected shoulder replacement. J Bone Joint Surg Br. 2008 Apr;90(4): 460-5.
- 9. Bauer TW, Parvizi J, Kobayashi N, Krebs V. Diagnosis of periprosthetic infection. J Bone Joint Surg Am. 2006 Apr;88(4):869-82.
- 10. Patel A, Calfee RP, Plante M, Fischer SA, Green A. Propionibacterium acnes colonization of the human shoulder. J Shoulder Elbow Surg. 2009 Nov-Dec;18 (6):897-902. Epub 2009 Apr 11.
- 11. Del Pozo JL, Patel R. Clinical practice. Infection associated with prosthetic joints. N Engl J Med. 2009 Aug 20;361(8):787-94.
- 12. Topolski MS, Chin PYK, Sperling JW, Cofield RH. Revision shoulder arthroplasty with positive intraoperative cultures: the value of preoperative studies and intraoperative histology. J Shoulder Elbow Surg. 2006 Jul-Aug;15(4):402-6.
- 13. Levy O, Iyer S, Atoun E, Peter N, Hous N, Cash D, Musa F, Narvani AA. Propionibacterium acnes: an underestimated etiology in the pathogenesis of osteoarthritis? J Shoulder Elbow Surg. 2013 Apr;22(4):505-11. Epub 2012 Sep 13.
- 14. Sch"afer P, Fink B, Sandow D, Margull A, Berger I, Frommelt L. Prolonged bacterial culture to identify late periprosthetic joint infection: a promising strategy. Clin Infect Dis. 2008 Dec 1;47(11):1403-9.
- 15. Dodson CC, Craig EV, Cordasco FA, Dines DM, Dines JS, Dicarlo E, Brause BD, Warren RF. Propionibacterium acnes infection after shoulder arthroplasty: a diagnostic challenge. J Shoulder Elbow Surg. 2010 Mar;19(2):303-7. Epub 2009 Nov 1.
- 16. Butler-Wu SM, Burns EM, Pottinger PS, Magaret AS, Rakeman JL, Matsen FA 3rd, Cookson BT. Optimization of periprosthetic culture for diagnosis of Propionibacterium acnes prosthetic joint infection. J Clin Microbiol. 2011 Jul;49(7):2490-5. Epub 2011 May 4.
- 17. Shannon SK, Mandrekar J, Gustafson DR, Rucinski SL, Dailey AL, Segner RE, Burman MK, Boelman KJ, Lynch DT, Rosenblatt JE, Patel R. Anaerobic thioglycolate broth culture for recovery of Propionibacterium acnes from shoulder tissue and fluid specimens. J Clin Microbiol. 2013 Feb;51(2):731-2.
- 18. Butler-Wu SM, Cookson BT. Reply to "Anaerobic thioglycolate broth culture for recovery of Propionibacterium acnes from shoulder tissue and fluid specimens". J Clin Microbiol. 2013 Feb;51(2):733.
- 19. Grosso MJ, Frangiamore SJ, Ricchetti ET, Bauer TW, Iannotti JP. Sensitivity of frozen section histology for identifying Propionibacterium acnes infections in revision shoulder arthroplasty. J Bone Joint Surg Am. 2014 Mar 19;96(6):442-7.
- 20. Frangiamore SJ, Saleh A, Kovac MF, Grosso MJ, Zhang X, Bauer TW, Daly TM, Ricchetti ET, Iannotti JP. Synovial fluid interleukin-6 as a predictor of periprosthetic shoulder infection. J Bone Joint Surg Am. 2015 Jan 7;97(1):63-70.

- 21. Grosso MJ, Sabesan VJ, Ho JC, Ricchetti ET, Iannotti JP. Reinfection rates after 1-stage revision shoulder arthroplasty for patients with unexpected positive intraoperative cultures. J Shoulder Elbow Surg. 2012 Jun;21(6):754-8. Epub 2012 Feb 3.
- 22. Kelly JD 2nd, Hobgood ER. Positive culture rate in revision shoulder arthroplasty. Clin Orthop Relat Res. 2009 Sep;467(9):2343-8. Epub 2009 May 12.
- 23. Ricchetti ET, Frangiamore SJ, Grosso MJ, Alolabi B, Saleh A, Bauer TW, Iannotti JP. Diagnosis of periprosthetic infection after shoulder arthroplasty: a critical analysis review. JBJS Reviews. 2013 Nov;1(1):e3.
- 24. Piper KE, Jacobson MJ, Cofield RH, Sperling JW, Sanchez-Sotelo J, Osmon DR, McDowell A, Patrick S, Steckelberg JM, Mandrekar JN, Fernandez Sampedro M, Patel R. Microbiologic diagnosis of prosthetic shoulder infection by use of implant sonication. J Clin Microbiol. 2009 Jun;47(6):1878-84. Epub 2009 Mar 4.
- 25. Nodzo SR, Hohman DW, Crane JK, Duquin TR. Hemolysis as a clinical marker for Propionibacterium acnes orthopedic infection. Am J Orthop (Belle Mead NJ). 2014 May;43(5):E93-7.